CLINICAL TRIAL: NCT01398176
Title: Immune Benefits From Mushroom Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MC-95320
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Humans
Keywords: gamma delta T cell; proliferation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 ounces of mushrooms (Experimental): 3 ounces of mushrooms consumed daily for 4 weeks
  Interventions: Dietary Supplement: 3 ounces of mushrooms
- 6 ounces of mushrooms (Experimental): 6 ounces of mushrooms consumed daily for 4 weeks
  Interventions: Dietary Supplement: 6 ounces of mushrooms

INTERVENTIONS:
Dietary Supplement: 3 ounces of mushrooms — 3 ounces of mushrooms consumed daily for 4 weeks
  Arms: 3 ounces of mushrooms
Dietary Supplement: 6 ounces of mushrooms — 6 ounces of mushrooms consumed daily for 4 weeks
  Arms: 6 ounces of mushrooms

SUMMARY:
The purpose of this study is to determine whether consuming mushrooms is effective in enhancing the function of γδ T cells.

DETAILED DESCRIPTION:
A non-therapeutic study is described. This is an intervention study at two levels of mushroom intake. The number of subjects and experimental assays are selected as a pilot study to generate the dose level and the efficacy. Subjects age 21 to 50 will be recruited and provide a baseline blood draw. The mushroom supplementation will occur for 4 weeks at two levels 85 g (3 ounces) and 170 g (6 ounces). Immunity changes fairly rapidly; in and early study the investigators saw changes in as little as 3 days. Blood is taken again at 4 weeks. Peripheral blood mononuclear cells are isolated from the blood and used freshly isolated, or cultured in autologous serum for 24 hours or for 10 days. Freshly isolated cells will be used to count γδ T cell and NK cells baseline values. After 24 hours of stimulation with a broad based mitogen, culture medium is harvested and assayed for cytokines secreted into the culture medium as well as NK cell activation and proliferation. Finally, cells are harvested after 10 days and assayed for γδ T cell activation and proliferation.

Consumers will benefit from knowing that health benefits can be derived from mushrooms. Potentially, this will stimulate mushroom sales and increase the variety of mushrooms consumed.

γδ T cells reside in epithelial linings of the lung, gut and reproductive tract and although their number is not precisely known, they are in much greater numbers than the circulating αβ T cells. γδ T cells are not activated in the same way as the αβ cells, they are activated more like cells of the innate immune system, by recognition of pathogen-associated molecular patterns (1,2). Recognition of pathogen-associated molecular patterns is rather non-specific, but very effective. For example, prenyl phosphate is a molecule having a pattern that is recognized by receptors of the γδ T cells. Interaction of prenyl phosphate with the γδ T cell receptor results in γδ T cell proliferation; expression of cell surface activation markers, such as cytokine receptors; and lastly, synthesis and secretion of cytokines necessary for communicating with other branches of the immune system. The investigators hypothesize that consuming mushrooms will result in greater proliferation when stimulated and will also enhance their capacity for activation, defined here as cytokine secretion and cell surface marker expression.

A second quality of γδ T cells is their ability to turn off the immune response once it is no longer needed. Carding and Egan (3,4) showed that γδ T cells were responsible for killing activated macrophages after the pathogen had been eliminated. Knockout mouse models show that the elimination of γδ cells promote chronic inflammation, prevent wound healing (5) and may increase the risk for cancer (6,7). The magnitude and the importance of the γδ T cell are just being realized. By strengthening γδ T cells, the investigators will fight pathogen better and resolve inflammation quicker.

It is our hypothesis that there are certain bioactive components that resemble pathogen-associated molecular patterns and interact weakly with the epithelial γδ T cells in such a way that they are "primed", but not activated. The bioactive food components do not interact with the cells with enough strength to cause an actual response, but, later, when the cells do encounter pathogen, they can react quicker and with more intensity if they have already been primed. The primary bioactive components in mushrooms that may interact with immune cells are polysaccharides and glycoproteins and the two major types of mushroom polysaccharides include glucans (both β and α) and heteroglycans. Additionally, mushrooms contain another important polysaccharide, chitin. Chitin is composed of N-acetyl-d-glucosamine units (8,9). These compounds are some likely candidates, in addition to other immuno-modulating compounds such as Vitamin D (10) and B vitamins.

Mushrooms have been shown to have an impact on immune cells, particularly NK cells (11,12) but the γδ T cell has not been studied. The composition of mushroom is well suited to interact with the γδ T cell. NK cell activity will be used in this study as a positive control although the investigators will use flow cytometry rather than generalized non-specific cytolytic activity.

The investigators know from our previous studies in humans (7,13,14) and from other published studies (15,16) that foods such as tea, apples, encapsulated fruits and vegetables contain compounds that appear to prime γδ T cells. The investigators hypothesize that bioactive compounds in the gut are recognized by intestinal γδ T cells, resulting in a primed cell. These cells are not static but migrate in and out of tissues, through the circulation as well as lymph nodes (17). Thus, the investigators can measure functional changes in the blood borne γδ T cells regardless of whether the bioactive compound is absorbed or not.

This study will specifically study the shiitake (Lentinus edodes) mushroom. This mushroom has been shown in other research to have a variety of health benefits, but few feeding trials, and none in healthy humans, has been done (18-20).

5. Specific Aims:

The aim is to determine if bioactive compounds in mushroom can enhance the activity of this cell type. Because this cell type resides in the epithelial linings and migrates via the blood and lymph system, the investigators can measure functional changes in this cell regardless of whether bioactive compounds are absorbed or not. It is often describe as the first line of defense.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female
* Between the ages of 21 and 50
* BMI between 18 and 35

Exclusion Criteria:

* Have illness at the time of enrollment
* On immunosuppressive drugs, antibiotics, chronic use of NSAIDS
* Ongoing infection or hypertension that requires medication
* Consume any flavonoid-containing supplements, antioxidant supplements or probiotics
* Consume more than 14 glasses of alcoholic beverages per week
* Consume more than 7 servings of fruits and vegetables per day
* Are on a strict vegetarian diet
* Pregnant or lactating women or individuals on hormone therapy

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Percival, PhD, Principal Investigator — University of Florida
Locations (1):
- 449 Food Science and Human Nutrition Department, Gainesville, Florida, United States

REFERENCES:
- [Derived] Dai X, Stanilka JM, Rowe CA, Esteves EA, Nieves C Jr, Spaiser SJ, Christman MC, Langkamp-Henken B, Percival SS. Consuming Lentinula edodes (Shiitake) Mushrooms Daily Improves Human Immunity: A Randomized Dietary Intervention in Healthy Young Adults. J Am Coll Nutr. 2015;34(6):478-87. doi: 10.1080/07315724.2014.950391. Epub 2015 Apr 11. PMID 25866155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in October 2011. Individuals responded to posted advertisements by calling. Eligibility was determined and the individual was assigned a time to come in for the first blood draw.
Pre-assignment Details: 52 participants were consented to the study; however, one participant who was consented was found to be in a conflicting study, and was dropped prior to the start of the study. 51 participants started the study interventions.
Period: Overall Study
Arm/Group | 3 Ounces of Mushrooms | 6 Ounces of Mushrooms
Started | 26 | 25
Completed | 23 | 19
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Ounces of Mushrooms | 6 Ounces of Mushrooms | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (2.14) | 25.6 (6.4) | 24.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Physiological Modifications to Gamma Delta T Cell Function
Description: Proliferation of γδ-T cells when cultured ex vivo in autologous serum. Values are expressed as a percent of CD3 cells, which means a percent of the total T cell population. Only T cells express CD3.
Time Frame: 4 weeks
Population: Intent to treat
Measure: Mean (Standard Error); unit: percent of T lymphocytes
Arm/Group | 3 Ounces of Mushrooms | 6 Ounces of Mushrooms
Number analyzed (Participants) | 26 | 25
percent of T lymphocytes | 22.65 (0.97) | 22.17 (1.01)

ADVERSE EVENTS:
Arm/Group | 3 Ounces of Mushrooms | 6 Ounces of Mushrooms
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

LIMITATIONS AND CAVEATS:
No specific limitations outside of the normal limitations to human interventions studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No